CLINICAL TRIAL: NCT01673152
Title: The Effect of the Oligofructose Supplementation on Body Weight in Overweight and Obese Children: a Randomized, Double Blind, Placebo-controlled Trial
Brief Title: The Effect of the Oligofructose Supplementation on Body Weight in Overweight and Obese Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: Nutricia Foundation (Other)
Responsible Party: Principal Investigator, Hanna Szajewska, Professor, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RG 4/2011
Record Dates: First submitted 2012-06-27; First posted 2012-08-27 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Obesity
Keywords: Obesity; Overweight; Satiety; Oligofructose; Prebiotic
MeSH Terms: conditions — Obesity; Overweight | interventions — oligofructose; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maltodextrin (Placebo Comparator)
  Interventions: Dietary Supplement: Maltodextrin
- Oligofructose (Experimental): Orafti P95, Beneo-Orafti, Belgium,
  Interventions: Dietary Supplement: Oligofructose

INTERVENTIONS:
Dietary Supplement: Oligofructose — Dosing: children aged 7 to 12 years: 8g/day, children aged 12 to18 years: 15g/day Duration: 12 weeks
  Other Names: Orafti P95, Beneo-Orafti, Belgium
  Arms: Oligofructose
Dietary Supplement: Maltodextrin — Dosing: children aged 7 to 12 years: 4g/day, children aged 12 to18 years: 6g/day, Duration: 12 weeks
  Arms: Maltodextrin

SUMMARY:
This study is designed to assess the effect of oligofructose administration for 12 weeks on Body Mass Index (BMI) of overweight and obese children.

DETAILED DESCRIPTION:
The prevalence of childhood overweight and obesity is reaching epidemic proportions. There have been no effective methods for preventing or treating obesity in childhood so far prompting interest in new interventions. One potential option for obesity prevention is the use of the prebiotic oligofructose. Data from research on rodents shows that a high-fat diet enriched with oligofructose causes a decrease in energy intake, less weight gain and a lower level of triglycerides . A similar effect has been observed in healthy adults. Available evidence suggests that the addition of oligofructose to the diets of overweight or obese adults may increase satiety and thus reduce energy intake. Currently, there are no data on the effect of oligofructose in overweight and obese children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7 to 18 years
* BMI > 85 percentile
* Signed informed consent

Exclusion Criteria:

* Overweight / obesity secondary to genetic syndromes and/or endocrine diseases

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 96 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
BMI z-score difference | after 12 weeks of the intervention

SECONDARY OUTCOMES:
BMI z-score difference | after 24 weeks of the intervention
Percentage of weight reduction | after 12 weeks of the intervention
Difference in total body fat measured by Dual-Energy X-ray Absorptiometry (DEXA) | after 12 weeks of the intervention
Percentage of children with BMI-for-age > 85percentile | after 12 and 24 weeks of the intervention
Mean BMI z-score | after 12 and 24 weeks of the intervention
Self-reported energy intake (3-day diet record) | after 12 weeks of the intervention
Percentage of the children with abnormal fasting glucose | after 12 weeks of the intervention
Percentage of the children with dyslipidemias | after 12 weeks of the intervention
Percentage of the children with hypertension | after 12 weeks of the intervention
Adverse effects | during intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Samodzielny Publiczny Dziecięcy Szpital Kliniczny, Warsaw, Poland